CLINICAL TRIAL: NCT04323241
Title: The Effect of Placenta Removal Method On Postpartum Leucocytosis : A Randomized Controlled Trial
Brief Title: Association of Placenta Removal Method and Postpartum Leucocytosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sevcan Arzu Arinkan, Medical Doctor, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HNEAH KAEK 2019/KK/10
Record Dates: First submitted 2020-03-05; First posted 2020-03-26 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Cesarean Section Complications
Keywords: Placenta removal method; postpartum leucocytosis; endometritis; postpartum anemia
MeSH Terms: conditions — Endometritis

STUDY DESIGN:
Intervention Model Description: The operative procedures are similar in all patients and followed the same technical steps. All patients are randomized according to the removal of placenta from the uterus after childbirth; manually removing placenta and control of endometrial cavity by fingers (Group 1) or controlled cord traction without putting fingers inside the uterus (Group 2).
Who Masked: Investigator
Masking Description: Investigator will not know the interventional group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): In group 1, plasenta is removed manually. Manual removal of the placenta will be performed by placing surgeon's dominant hand in the uterine cavity and removing the placenta by detaching it from the uterine wall as soon as possible after the delivery of the infant. The emptiness of the uterine cavity is verified manually.
- Study Group (Experimental): In group 2, plasenta is removed by controlled cord traction. Spontaneous removal will be performed by external uterine massage and traction on the umbilical cord are performed to assist spontaneous delivery of the placenta.
  Interventions: Other: Controlled cord traction

INTERVENTIONS:
Other: Controlled cord traction — In group 2, Spontaneous removal will be performed by massaging on the uterine fundus and applying gentle traction on the umbilical cord.
  Arms: Study Group

SUMMARY:
Cesarean delivery is one of the most common major abdominal operation in women worldwide. The incidence of postpartum infection has been estimated to be 1-4% after vaginal delivery and 10-20% after Cesarean delivery. Although it is widely performed, manual removal of the placenta is still a conflicting issue due to the risk of post-partum endometritis. All cesarean patients are randomized according to the removal of placenta from the uterus after childbirth; manually (Group 1) or controlled cord traction without putting fingers inside the uterus (Group 2). The aim of this study is to examine whether there is an association between the method of removal of the placenta and postpartum white blood cell increase in nonanemic, singleton, low-risk group of women with term pregnancies, who underwent elective cesarean delivery under general anesthesia.

DETAILED DESCRIPTION:
Objective:

Cesarean section is one of the most common major abdominal operation in women worldwide and its rate is increasing every year. Although cesarean birth is considered as safe, it is a potentially morbid procedure with associated risks of hemorrhage, thromboembolic events, infection, and anesthesia risks. The incidence of postpartum infection has been estimated to be 1-4% after vaginal delivery and 10-20% after cesarean section. Manual removal of the placenta is widely accepted by surgeons worldwide. This method enables the surgeon quick intervention. Beside, it helps uterine cavity to be examined for damage and the presence of placental remnants. However, manual removal of the placenta is still a conflicting issue due to the risk of post-partum endometritis, post-partum hemorrhage and abnormal placentation in subsequent pregnancies. It is assumed that controlled cord traction reduces the risk of postpartum hemorrhage and infection.

The aim of this study is to examine whether there is an association between the method of removal of the placenta and increase in postpartum white blood cell counts

After informed consent, all patients are randomized according to the removal of placenta from the uterus after childbirth; manually (Group 1) or controlled cord traction without putting hands inside the uterus (Group 2). Patients are examined regarding to maternal infection. BMI measurement, obstetrics and medical history are recorded. The operative procedures are similar in all patients and followed the same technical steps. In both groups, oxytocin and a first-generation cephalosporin antibiotic are administered intravenously after the delivery of the infant. All uterine incisions were low transverse and all were closed without exteriorisation of the uterus. Complete blood count before delivery, on pastpartum day 1 and 2, fever during hospitalisation, average blood loss during operation and the endometritis cases are recorded. All the patients are asked to come to control on postpartum day 10. Also, patients are asked to come to control if they have fever, abnormal vaginal bleeding, abnormal vaginal discharge, general feeling of sickness and pain in the pelvis. Fever is defined as a temperature above 38.5°C on two consecutive days, excluding the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Nonanemic pregnancies
* Singleton pregnancies
* Term pregnancies
* Elective cesarean sections

Exclusion Criteria:

* Patients having umbilical cord prolapse,
* Patients having placenta previa
* Patients having preterm rupture of mebranes
* Patients having maternal infection
* Patients having multiple gestation
* Patients having antepartum hemorrhage
* Patients having severe pre-eclampsia
* Patients having placenta previa
* Patients having placental abruption
* Patients having uncontrolled gestational diabetes
* Heart disease
* Liver disorders
* Renal disorders
* Coagulopathy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Leukocyte Level at Postpartum Day 1 | Before delivery and postpartum day 1
  Measurement of complete blood count
Detection of Leukocyte Count | Postpartum day 2
  Measurement of complete blood count
Detection of Number of Patients with Fever | On postpartum day 1
  Body temperature is measured 4 times in a day. Highest temparature will be record on postpartum day 1.
Detection of Number of Patients with Fever | On postpartum day 2
  Body temperature is measured 4 times in a day. Highest temparature will be record on postpartum day 2.
Number of Participants with Postpartum Endometritis | Postpartum day 10
  All the patients are asked to come to control on postpartum day 7. Also, patients are asked to come to control if they have fever, abnormal vaginal bleeding, abnormal vaginal discharge, general feeling of sickness and pain in the pelvis.

SECONDARY OUTCOMES:
Measurement of average blood loss during caesarean section by change from baseline hematocrit level at postpartum day 1. | Before operation and postpartum day 1
  Measurement of hematocrit level

CONTACTS AND LOCATIONS:
Overall Officials: Sevcan Arzu Arinkan, M.D., Principal Investigator — Haydarpasa Numune Training and Research Hospital
Locations (1):
- University of Health Sciences Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT04323241/Prot_SAP_000.pdf